CLINICAL TRIAL: NCT01822028
Title: A Single-center, Double-blind, Randomized, Placebo-controlled, Two Period / Two Treatment Cross-over Study to Assess the Effect of Florastor® (Saccharomyces Boulardii Lyo) on Gastrointestinal Tolerability, Safety, and Pharmacokinetics of Zavesca® (Miglustat) in Healthy Subjects
Brief Title: Two Period / Two Treatment Cross-over to Assess the Effect of Florastor® on Gastrointestinal Tolerability, Safety, and PK in Healthy Subjects Receiving Zavesca®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AC-056-102
Record Dates: First submitted 2013-03-06; First posted 2013-04-02 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Diarrhea
Keywords: diarrhea
MeSH Terms: conditions — Diarrhea | interventions — miglustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Placebo Comparator): Treatment A: Florastor® 500 mg twice per day from Day 1 to Day 16 of the treatment period, and Zavesca® 100 mg three times per day from Day 3 to Day 16.
  For Period 2, subjects will receive the alternate dosing regimen.
  Interventions: Drug: Treatment A; Drug: Treatment B
- Treatment B (Experimental): Treatment B: Florastor® 500 mg twice per day from Day 1 to Day 16 of the treatment period, and Zavesca® 100 mg three times per day from Day 3 to Day 16.
  For Period 2, subjects will receive the alternate dosing regimen.
  Interventions: Drug: Treatment A; Drug: Treatment B

INTERVENTIONS:
Drug: Treatment A — Florastor® placebo. Zavesca® capsules dosed at 300 mg daily (one 100 mg capsule three times per day).
  Other Names: Florastor® placebo.; Zavesca® capsules.
Drug: Treatment B — Florastor® capsules dosed at 1000 mg daily (two 250 mg capsules two times per day).
  Zavesca® capsules dosed at 300 mg daily (one 100 mg capsule three times per day).
  Other Names: Florastor® capsules.; Zavesca® capsules.

SUMMARY:
Cross-over, tolerability study with healthy subjects taking Zavesca in combination with Florastor. Forty-two subjects will be randomized to one of two treatment sequences of Zavesca with Florastor and Zavesca with Placebo of Florastor. Gastrointestinal tolerability and PK endpoints, demographic, laboratory and safety testing, and AEs and SAEs will be collected throughout the seventy-four day study.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, double-blind, randomized, placebo-controlled, two period / two treatment, cross-over study with GI tolerability, safety, and PK assessments. A total of 42 healthy subjects will be enrolled. At least 30% of female subjects are expected to be enrolled. Subjects will participate in 2 treatment periods (Treatment Period 1 and Treatment Period 2), separated by a 10- to 14-day washout.

Subjects will be randomly allocated to the treatment sequence, A-B or B-A:

* Treatment A: Placebo of S. boulardii 500 mg twice a day (b.i.d.) from Day 1 to Day 16 of the treatment period, and miglustat capsules 100 mg t.i.d. from Day 3 to Day 16.
* Treatment B: S. boulardii 500 mg b.i.d. from Day 1 to Day 16 of the treatment period, and miglustat capsules 100 mg t.i.d. from Day 3 to Day 16.

To minimize possible carry-over effect, a 10 to 14-day washout period is added between Treatment Period 1 and Period 2. Steady-state PK evaluations will occur at the end of Period 1 and Period 2 requiring full-day clinic stays by each subject.

The planned study duration per subject will be approximately 46 days (not inclusive of Screening and serious adverse event [SAE] follow-up periods). However, the duration may be up to 53 days if all visit windows are utilized. The Screening period may last up to 30 days prior to the first administration of study medication. Telephone follow-up will occur within 48-72 hours after last study drug dose in each treatment period to record SAEs/AEs and concomitant medications. In addition, subjects will be followed up 30 days after permanent study drug discontinuation for ongoing AEs and new SAEs via a telephone consult.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* Healthy male and female subjects aged between 18 and 55 years (inclusive) at Screening
* Women must have a negative serum pregnancy test at Screening and negative urine pregnancy test at the first day of each treatment period and must use a reliable method of contraception from Screening during the entire study and up to 30 days after the last dose. Male subjects must agree to use reliable contraception throughout the study and for 4 months after study drug discontinuation
* Reliable methods of contraception for all subjects include the following:
* Barrier type devices (e.g., male and female condom, diaphragm and contraceptive sponges) used ONLY in combination with a spermicide
* Intrauterine devices
* Oral contraceptive agent
* Depo-Provera (medroxyprogesterone acetate)
* Levonorgestrel implants
* Abstinence, the rhythm method, and contraception by the partner alone are NOT reliable methods of contraception
* A BMI of 18.5 to 30 kg/m2 (inclusive) at Screening
* No clinically significant findings on the physical examination, laboratory assessment, electrocardiogram (ECG), and vital signs at Screening

Exclusion Criteria:

* Ingestion of any medication within 7 days prior to study enrollment (Day 1) except contraceptives
* Use of anti-diarrheal medications within 30 days prior to study enrollment (e.g., loperamide)
* Use of oral probiotic supplements or S. boulardii within 30 days prior to study enrollment
* Use of oral antifungals or antibiotics within 8 weeks prior to study enrollment
* History of yeast allergy
* Current alcohol or drug dependence
* Renal function impairment, (i.e., creatinine clearance [C Cr]<70 mL/min/1.73m2 as per Cockroft-Gault)
* History of GI distress including diarrhea (more than 2 loose stools per day, for 5 or more days) within 30 days prior to study enrollment
* History of irritable bowel syndrome, inflammatory bowel disease, or other disease resulting in frequent or severe diarrhea
* Lactose intolerance
* Subjects on any specialized diet, including low carbohydrate diets Lactating, pregnant women or women who plan to become pregnant during the course of the study
* History of any neurological disease/symptom, e.g., convulsion
* Loss of 500 mL or more of blood within 3 months prior to Screening
* Positive results to HIV Ag/Ab, HBsAg or anti-HCV tests
* Positive results from the HIV serology at Screening
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to Screening
* Excessive caffeine consumption, defined as >=5 cups of coffee a day or 800mg/day at Screening
* Smoking within 3 months prior to Screening and inability to refrain from smoking during the course of the study
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol
* Legal incapacity or limited legal capacity at Screening
* Unplanned weight loss defined as >5% within the past month or >=10% during the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
GASTROINTESTINAL TOLERABILITY ENDPOINTS | baseline to end of study (day 74)
  Total number of days of diarrhea defined as 3 or more loose stools within a 24-hour period (WHO criteria) that meet the criteria of Bristol Stool Score 6-7.

SECONDARY OUTCOMES:
GASTROINTESTINAL TOLERABILITY ENDPOINTS | baseline to end of study (day 74)
  Number of consecutive days of diarrhea defined as 3 or more loose stools (WHO criteria) within consecutive 24-hour periods that meet the criteria of Bristol Stool Score of 6-7.

OTHER OUTCOMES:
PHARMACOKINETIC ENDPOINTS | day 16 and day 44
  Plasma PK parameters will be derived by non-compartmental analysis of the concentration-time profiles of miglustat following the last dose at end of Periods 1 and 2. The area under the plasma concentration-time curve during a dosing interval (AUCt). The maximum plasma concentration (Cmax). The time to reach maximum plasma concentration (tmax).
GENERAL TOLERABILITY/SAFETY ENDPOINTS, OTHER THAN GASTRO-INTESTINAL EVENTS | baseline to end of study (day 74)
  Treatment-emergent adverse events (TEAEs) up to 48 hours after the last study drug dose in each treatment period. Leading to the premature discontinuation of study drug. Treatment-emergent SAEs up to 48 hours after the last study drug dose in each treatment period. Change from baseline to EOT in body weight and vital signs blood pressure (BP) and heart rate (HR).

CONTACTS AND LOCATIONS:
Overall Officials: Chad McQueen, PharmD, Study Director — Actelion
Locations (1):
- BioPharma Services Inc., Toronto, Ontario, Canada